CLINICAL TRIAL: NCT02907996
Title: A Post-Marketing Surveillance Study to Evaluate the Safety and Effectiveness of Sovaldi in Patients With Chronic Hepatitis C Virus (HCV) Infection in Korea
Brief Title: Evaluate the Safety and Effectiveness of Sovaldi in Participants With Chronic Hepatitis C Virus (HCV) Infection in Korea
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-334-1967
Record Dates: First submitted 2016-09-16; First posted 2016-09-20 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sofosbuvir: Adult Korean participants with genotype 1, 2, 3, and 4 chronic HCV infection and pediatric Korean participants aged 12 to <18 years with genotype 2 and 3 chronic HCV infection who are initiating commercial Sovaldi regimens
  Interventions: Drug: Sofosbuvir

INTERVENTIONS:
Drug: Sofosbuvir — 400 mg tablet administered orally once daily
  Other Names: Sovaldi ®

SUMMARY:
The objectives of this study are to collect and assess data related to safety and effectiveness of Sovaldi treatment regimens, per the approved prescribing information for Sovaldi, in routine clinical practice and report results to Korean Ministry of Food and Drug Safety (MFDS).

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals aged 12 years and older who are living in Korea
* Individuals with chronic HCV infection eligible for treatment with Sovaldi as indicated in the approved prescribing information for Sovaldi
* Individuals who have been informed of all pertinent aspects of the study and have voluntarily signed Personal Information Protection Act (PIPA) consent form; Pediatric individuals who have their legally authorized representatives sign the PIPA consent form

Key Exclusion Criteria:

* Individuals treated with Sovaldi outside of the approved prescribing information for Sovaldi in Korea
* Individuals who have a contra-indication (refer to the Korea prescribing information)
* Individuals who have a contra-indication to ribavirin or peginterferon alfa or daclatasvir
* Pregnant or breast feeding women
* Individuals who have previously been administered Sovaldi
* Individuals participating in a concurrent HCV clinical trial
* Individuals planning on leaving the country during the study period

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult Korean individuals with Genotype 1, 2, 3, and 4 chronic HCV infection and pediatric Korean individuals (aged 12 to <18 years) with genotype 2 and 3 chronic HCV infection who are initiating commercial Sovaldi regimens.
Sampling Method: Non-Probability Sample
Enrollment: 2033 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Any Adverse Events (AEs) Occurring During Administration of Sovaldi Regimens or Within 30 Days After Completion (or Discontinuation) of Sovaldi Treatment Regimens | First dose date up to 30 days posttreatment
Proportion of Participants with HCV RNA < Lower Limit of Quantification (LLOQ) | 2 weeks before Posttreatment Week 12 through Week 24 Posttreatment

SECONDARY OUTCOMES:
Percentage of Participants Experiencing Any AEs Occurring During Administration of Sovaldi Regimens or Within 12 Weeks After Completion (or Discontinuation) of Sovaldi Treatment Regimens | First dose date up to 12 weeks posttreatment

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (71):
- South Korea (71):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - CHA Bundang Medical Center, Sungnam, Gyeonggi-d
  - Hallym University Sacred Heart Hospital, Anyang
  - The Catholic University of Korea Bucheon ST. Mary's Hospital, Bucheon-si
  - SoonChunHyang University Bucheon Hospital, Bucheon-si
  - Inje University Haeundae Paik Hospital, Busan
  - BongSeng Memorial Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Busan St. Mary's Hospital, Busan
  - Busan Veterans Hospital, Busan
  - Maryknoll Medical Center, Busan
  - Changwon Fatima Hospital, Changwon
  - Dankook University Hospital, Cheonan
  - SoonChunHyang University Cheonan Hospital, Cheonan
  - Hallym University ChunCheon Sacred Heart Hospital, Chuncheon
  - Konkuk University Chungju Hospital, Chungju
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Kyungpook national university medical center Chil-Gok, Daegu
  - DaeJeon ST. Mary's Hospital, Daejeon
  - Chungnam National University Hospital, Daejeon
  - Daejeon Eulji Medical Center, Daejeon
  - GangNeung Asan Hospital, Gangneung
  - Dongguk University Ilsan Hospital, Goyang
  - Myongji Hospital, Goyang
  - National Health Insurance Cooperation Ilsan Hospital, Goyang-si
  - Kumi Cha Hospital, Gumi
  - Hanyang University Guri Hospital, Guri-si
  - Konkuk University Medical Center, Gwangjin-gu
  - Chosun University Hospital, Gwangju
  - Kwangju Christian Hospital, Gwangju
  - Dongguk University Gyeongju Hospital, Gyeongju
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Chonnam National University Hwasun Hospital, Hwasun
  - WonKwang University Hospital, Iksan
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Inha University Hospital, Incheon
  - Catholic Kwandong University International St. Mary's Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Cheju Halla General Hospital, Jeju City
  - Presbyterian Medical Center, Jeonju
  - Chonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - SoonChunHyang University Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Boramae Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Inje University Seoul Paik Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Nowon Eulji Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - The Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan
  - Yongin Severance Hospital, Yŏngin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-334-1967